CLINICAL TRIAL: NCT00277836
Title: A Phase 1 Dose-Escalation Study of Intravenous MST-997 Formulated in Polysorbate 80 Diluent Administered Weekly in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating MST-997 in Advanced Malignant Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 3161K1-101
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2006-12-08 (Estimated); Status verified 2006-12

CONDITIONS: Neoplasms
Keywords: malignant tumor
MeSH Terms: conditions — Neoplasms | interventions — MST 997

INTERVENTIONS:
Drug: MST-997

SUMMARY:
MST-997 is a taxane analog with the potential to treat subjects with a variety of tumor types. Preclinical data demonstrated that MST-997 inhibited tumor growth when administered intravenously (IV). This phase 1 dose escalation study is designed to evaluate the safety and tolerability of if IV MST-997 formulated in Polysorbate 80 Diluent can be safely administered on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of malignant solid tumor with measurable disease
* Life expectancy of at least 12 weeks
* ECOG (Eastern Cooperative Oncology Group) performance status of 0,1,or 2

Exclusion Criteria:

* Recent major surgery, radiation therapy or anti-cancer treatment
* History of any other prior malignancy within last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

PRIMARY OUTCOMES:
To evaluate the safety, tolerability and MTD (maximum tolerated dose) of MST-997.

SECONDARY OUTCOMES:
Preliminary pharmacokinetic information on the pharmacokinetics (during cycle 1) abd anti-tumor activity (assessed approximately every 8 weeks) of on MST-997

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Poland, WPWZMED@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com
Locations (1):
- Houston, Texas, United States